CLINICAL TRIAL: NCT03073135
Title: Randomized Controlled Trial of Group Psychodrama for Skin Picking
Brief Title: Group Psychodrama for Skin Picking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Hermano Tavares, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #14760
Record Dates: First submitted 2016-04-29; First posted 2017-03-08 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Excoriation of Skin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychodrama Group Therapy (PGT) (Experimental): The PGT is a 15-session weekly program. Sessions last one and a half hours, conducted by two psychologists with more than ten years of experience. The process will be divided into three stages: the first (5 sessions) will be focused on the management of the individual's relationship challenges. The second stage (5 sessions) will focus on the association between the subject's management of their relationships and the excoriation disorder (ED) symptoms. The third (5 sessions) will focus on the development of new skills for the management of ED. Psychodramatic methods will be used throughout the process.
  Interventions: Behavioral: Psychodrama Group Therapy (PGT)
- Supportive Group Therapy (SGT) (Active Comparator): The SGT is a 15-session weekly program. Sessions last one and a half hours, conducted by two psychologists with more than ten years of experience.
  Interventions: Behavioral: Supportive Group Therapy (SGT)

INTERVENTIONS:
Behavioral: Psychodrama Group Therapy (PGT) — The psychotherapeutic focus is on the "here and now" aspect of the patient's relationships. Conflicts are acted out during the sessions, yielding intense emotional re-experience in a safe environment, which will bring further cognitive understanding of past distressful life experiences and hopefully new adaptive ways of expressing and dealing with the problem.
  Arms: Psychodrama Group Therapy (PGT)
Behavioral: Supportive Group Therapy (SGT) — SGT is a form of treatment in which the therapist maintains a therapeutic relationship and a working alliance based on reality, support, clarification, assistance in troubleshooting, strong leadership, partial gratification of dependency needs, legitimating independence, development of pleasurable activities and adequate rest, guidance and advice to deal with current problems. This approach uses techniques to help patients feel safe, accepted, protected, encouraged and not anxious.
  Arms: Supportive Group Therapy (SGT)

SUMMARY:
This study aims to evaluate the effectiveness of psychodrama group therapy (PGT) compared with supportive group therapy (SGT) for excoriation disorder (ED). Patients will be randomly allocated for either PGT or SGT. The Skin Picking Scale Revised (SPS-R) will be the primary outcome and emotional regulation measured by the Difficulties in Emotion Regulation Scale (DERS) will be evaluated as a potential intermediator. The Clinical Global Impression Scale (CGI); Beck Depression Scale (BDI); Beck Anxiety Scale (BAI), and the Social Adjustment Scale (EAS) will assess secondary outcomes.

DETAILED DESCRIPTION:
Excoriation disorder (ED) is a diagnostic characterized by recurrent picking at one´s own skin, resulting in skin lesions, despite repeated attempts to stop the behavior that causes clinically significant distress or impairment in important areas of functioning. The skin picking behavior is better accounted by physiological effects of a substance or better explained by symptoms of another mental disorder.

Objective: This study aims to evaluate the effectiveness of psychodrama group therapy (PGT) compared with supportive group therapy (SGT).

Justification: The scientific studies on treatment for ED are scarce and all associated with behavioral therapy methods, which do not adequately consider underlying factors of ED, such as emotional dysregulation. There are also not reports of group treatment for ED.

Method: patients who meet criteria for ED according to DSM-5 will be selected . Patients in need of treatment for psychiatric comorbidities (such as anxiety and depression) will wait at least 4 weeks until pharmacological prescription is stable. The subjects will be randomly allocated to either PGT or SGT. The Skin Picking Scale Revised (SPS-R) will be the primary outcome and emotional regulation measured by the Difficulties in Emotion Regulation Scale (DERS) will be evaluated as a potential intermediator. The Clinical Global Impression Scale (CGI); Beck Depression Scale (BDI); Beck Anxiety Scale (BAI), and the Social Adjustment Scale (EAS) will assess secondary outcomes.

Hypotheses:

1. The PGT is more effective than SGT for the ED patient regarding the reduction of skin excoriation behavior.
2. PGT is more effective than SGT for the ED patient regarding the improvement of the symptoms of anxiety, depression and trichotillomania (when present).
3. The therapeutic effects of PGT is intermediated by emotional regulation.

ELIGIBILITY:
Inclusion Criteria:

* Skin Picking diagnosis

Exclusion Criteria:

* Illiteracy
* Other acute psychiatric diagnosis in need of inpatient treatment
* Mental retardation
* Prader-Willi syndrome or other medical condition causing recurrent excoriation behavior or intense itching

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Skin Picking Scale Change | Baseline, week 5, week 10, week 15
  Self-report questionnaire

SECONDARY OUTCOMES:
Difficulties in Emotion Regulation Scale Change | Baseline, week 5, week 10, week 15.
  Self-report questionnaire

OTHER OUTCOMES:
The Clinical Global Impression Scale Change | Baseline, week 15 (end of treatment.).
  semi structured interview with psychiatrist
Beck Depression Scale Change | Baseline, week 15 (end of treatment.).
  Self-report questionnaire
Beck Anxiety Scale Change | Baseline, week 15 (end of treatment.).
  Self-report questionnaire
Social Adjustment Scale Change | Baseline, week 15 (end of treatment.).
  Self-report questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da faculdade de medicina da Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No